CLINICAL TRIAL: NCT04216927
Title: Efficacy of Nitric Oxide Administration During Cardiopulmonary Bypass in Neonates at Reducing the Risk of Acute Kidney Injury
Brief Title: NO During CPB in Neonates to Reduce Risk of AKI
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Mallinckrodt (Industry); Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: MOD00004808
Record Dates: First submitted 2019-12-04; First posted 2020-01-03 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: AKI; CHD - Congenital Heart Disease; Surgery
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Nitric Oxide; Oxygen

STUDY DESIGN:
Intervention Model Description: • This pilot study is a single center, double-blind, randomized controlled trial.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Nitric Oxide (Experimental): Intraoperative NO entrained at 20 ppm into the oxygenator of the CPB circuit with standard care
  Interventions: Drug: Nitric Oxide
- Oxygen (Placebo Comparator): Standard CPB without NO administered at any point intraoperatively
  Interventions: Drug: Oxygen

INTERVENTIONS:
Drug: Nitric Oxide — gNO will be entrained at 20 ppm into the oxygenator of the CPB circuit
  Arms: Nitric Oxide
Drug: Oxygen — Oxygen alone will be entrained for placebo arm
  Arms: Oxygen

SUMMARY:
Acute kidney injury (AKI) following cardiac surgery for congenital heart defects (CHD) in children affects up to 60% of high risk-patients and is a major cause of both short- and long-term morbidity and mortality. Despite effort, to date, no successful therapeutic agent has gained widespread success in preventing this postoperative decline in renal function. Nitric oxide is an intricate regulator of acute inflammation and coagulation and is a potent vasodilator. The investigators hypothesize that nitric oxide, administered during cardiopulmonary bypass (CPB), may reduce the incidence of AKI.

ELIGIBILITY:
Inclusion Criteria:

* All neonates (≤31 days) undergoing cardiac surgery with CPB for CHD will be deemed eligible for enrollment.

Exclusion Criteria:

1. Failure to obtain informed consent from parent/guardian
2. Clinical signs of preoperative persistent elevated pulmonary vascular resistance,
3. Emergency surgery,
4. Episode of cardiac arrest within 1 week before surgery,
5. Recent treatment with steroids and/or a condition that may require treatment with steroids (excluding steroid administration specifically for CPB),
6. Use of inhaled NO (iNO) immediately prior to surgery,
7. Structural renal abnormalities by ultrasound,
8. Preoperative AKI,
9. Use of other investigational drugs,
10. Weight less than <2 kg,
11. Gestational age <36 weeks,
12. Major extracardiac congenital anomalies,
13. Non-English speakers.

Ages: 1 Day to 31 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
AKI | 72 hours
  Incidence of AKI in the first 72 hours postoperative as defined by the Kidney Disease Improving Global Outcomes (KDIGO) diagnostic classification

SECONDARY OUTCOMES:
Biomarker evidence of AKI - NGAL | 72 hours
  Incidence of structural AKI in the first 72 hours postoperative will be assessed by measurement of urine biomarker neutrophil gelatinase-associated lipocalin (NGAL)
Biomarker evidence of AKI - KIM-1 | 72 hours
  Incidence of structural AKI in the first 72 hours postoperative will be assessed by measurement of urine biomarker kidney injury molecule-1 (KIM-1)
Biomarker evidence of AKI - IL-18 | 72 hours
  Incidence of structural AKI in the first 72 hours postoperative will be assessed by measurement of urine biomarker interleukin-18 (IL-18)
Biomarker evidence of AKI - L-FABP | 72 hours
  Incidence of structural AKI in the first 72 hours postoperative will be assessed by measurement of urine biomarker liver-type fatty acid-binding protein (L-FABP)
Biomarker evidence of AKI - urinary nitrite | 72 hours
  Incidence of structural AKI in the first 72 hours postoperative will be assessed by measurement of urine biomarker urinary nitrate.
Impact on GFR | 72 hours
  Postoperative GFR measured using serum cystatin C.
Low Cardiac Output | 48 hours
  Incidence of low cardiac output syndrome (LCOS) during the first 48 hours postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No